CLINICAL TRIAL: NCT06442826
Title: Efficacy of Non-invasive Auricular Simulation for Exam Anxiety and Depression in University Students: A Pilot 3-arm Randomised Controlled Trial
Brief Title: Non-invasive Auricular Simulation for Exam Anxiety and Depression in University Students
Acronym: AURITEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Tecnocampus Mataró-Maresme (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 8/2023
Record Dates: First submitted 2024-05-30; First posted 2024-06-04 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-06

CONDITIONS: Anxiety; Stress; Insomnia
MeSH Terms: conditions — Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- True non-invasive auricular stimulation (TniAS) (Experimental): Ear stimulation using true ear patches
  Interventions: Other: Non-invasive auricular stimulation
- Sham auricular stimulation (SAS) (Placebo Comparator): Ear stimulation using sham ear patches
  Interventions: Other: Sham auricular stimulation (SAS)
- No-intervention group (NI) (No Intervention): Participants in the No-Intervention group (NI) will not receive any active intervention as part of the trial.

INTERVENTIONS:
Other: Non-invasive auricular stimulation — Single session TniAS stimulation will be achieved by applying four stimulation patches. These patches consist of stainless steel spheres with a diameter of 1.2 mm, covered with adhesive circular paper measuring 8 mm in diameter.
  Point 1. Located in the Triangular Fossa, upper and central level at the vertex of the Fossa, at junction between the upper root and the lower root of the Antihelix.
  Point 2. Located in the inner part of the Cymba (upper) conchae, in the angle formed by the lower root of the antihelix and the ascending branch of the Helix.
  Point 3. Located in the middle depression of the Cavum (lower) conchae.
  Poinit 4. It is located at the inner superior quadrant of Lobe, below the external curve of the Intertragus notch, in a depression 3-4 mm from the insertion of the lobe to the face.
  Arms: True non-invasive auricular stimulation (TniAS)
Other: Sham auricular stimulation (SAS) — Sham intervention will be conducted following the exact same procedure as the TniAS group, with the only difference being the use of sham stimulation patches. These sham patches will consist of the same patches utilized in the TniAS group, except for the absence of the stainless steel spheres. During the application of these sham patches, the investigator will adhere to the identical process as in the TniAS group, with the exception that no palpation will be performed to locate the exact points, and only minimal pressure required for patch adherence will be applied to minimize any substantial stimulation. Participants in the SAS group will also be explicitly instructed not to stimulate the points until the removal of the patches.
  The removal of the sham stimulation patches will follow the precise protocol applied in the TniAS group, ensuring consistency in the study procedures across both groups.
  Arms: Sham auricular stimulation (SAS)

SUMMARY:
In Spain, depression, anxiety, and stress are highly prevalent in the general population as well as in college students. In college students, Ramón Arbués et al. found a moderate prevalence of depression (18.4%), anxiety (23.6%) and stress (34.5%). It is essential to take responsibility for promoting health education, disease prevention, protection and care for young people.

Academic performance can be altered due to the stressful nature of exam situations, which can lead to increased anxiety and decrease expected performance, mainly due to effects such as decreased attention span, concentration and retention of information.

Modulation of vagal tone is a therapeutical strategy to heightened parasympathetic activity and withdrawal sympathetic activity. Auricular transcutaneous VNS (ATVNS) by which parasympathetic nerve system is modulated by means of the stimulation of the auricular branch of the vagus nerve that provides somatosensory innervation to the external ear.

It has been shown that there are different effective interventions to reduce the symptoms of stress, depression, anxiety and insomnia in university students, but they are based on psychological interventions or face-to-face and cognitive-behavioral therapeutic approach, so this study proposal incorporates noninvasive atrial stimulation as an alternative to traditional treatments, which apart from being cost-effective, is easy to apply, well tolerated and presumably can have beneficial effects in the short term.

In the present pilot study, authors propose to investigate the degree of depression, anxiety and stress on crucial dates of final exams of 1st year students of the Double Degree Physiotherapy - Physical Activity and Sport Sciences of the Health Department of the TecnoCampus.

Investigators will also evaluate the feasibility of a study to assess the efficacy of a non-pharmacological intervention, through a neuroreflex stimulation of vagal tone, with a non-invasive atrial stimulation protocol.

DETAILED DESCRIPTION:
Personal pronouns have been removed

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Tecnocampus undergraduate students from Physical Therapy and Sports Science Double Degree of 1rst course.
* To sign the informed consent
* Understand Catalan or Spanish language
* With the intention to attend to the first call exams of the 2nd trimester.

Exclusion Criteria:

* Receiving pharmacological medication for anxiety or mental disorders
* Receiving psychological treatment
* Pregnancy or breastfeeding
* Participants with part-time enrolment
* With skin lesions in both auricula,
* Participating in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Recruitment strategy effectiveness | Week 0
  o evaluate the effectiveness of our recruitment strategy, we will analyze several key metrics, including the number of eligible participants, the number who expressed interest by completing the initial form, the participants who proceeded to the initial interview, and finally, the number of students who enrolled in the study. Additionally, we will carefully examine the reasons provided by students who declined to participate, allowing us to refine our recruitment approach.
Safety and Tolerability | Week 2
  Any side effects that may arise during the study will be meticulously monitored, and their frequency and severity will be assessed based on patients' self-reports. These side effects will be categorized as either minor, relevant, or important according to the patients' descriptions and assessments. Additionally, we will maintain a record of the number of participants who chose to remove at least one of the patches due to the side effects they experienced

SECONDARY OUTCOMES:
Exclusion rate | Week 0
  The exclusion rate will be analyzed based on the percentage of participants interested in the study who do not fulfill the inclusion criteria. Additionally, reasons for exclusion will be documented.
Dropout rate | Week 2
  We will meticulously record and analyze the percentage of participants who discontinue or withdraw from the study, which means they do not attend the final assessment session. Detailed information about the reasons for dropout will be collected to gain valuable insights into participant retention and engagement throughout the study
Compliance to the intervention protocol | Week 2
  We will assess the percentage of participants who adhere to the treatment protocol. Participants will be considered adherent if at least two out of the four auricular stimulation patches remain in place at the final assessment visit. Adherence will be evaluated based on self-reported information provided by participants during the last assessment interview.
Data collection feasibility | Week 2
  We will evaluate the feasibility of our data collection methods by gauging participants' perceptions of the ease of administration, comprehensibility, and time required for data collection. This assessment will employ a 5-point Likert scale and will be complemented by qualitative feedback. Additionally, outcome assessors will record any difficulties encountered during the data collection process.
Participant blinding success: | Week 2
  To determine the success of participant blinding, we will inquire during the final assessment session whether participants believe they received an active treatment. They will be provided with response options including "Yes," "No," or "I don't know.
Outcome assessor blinding success | Week 2
  he success of outcome assessor blinding will be assessed at the end of the final evaluation of each participant. Assessors will have to choose between 3 possible answers; "the participant was in the intervention group", "the participant was in the sham group", or "I don't know".
Anxiety | Week 2
  We will employ the DASS anxiety subscale to measure participants' anxiety levels. This subscale comprises questions that delve into anxiety-related feelings and experiences, providing a quantitative measure of anxiety symptomatology. Higher scores on this subscale indicate greater levels of anxiety.
Stress | Week 2
  The DASS instrument includes a stress subscale that helps us assess participants' stress levels. Participants will respond to items that reflect stress-related experiences, allowing us to quantify their perceived stress. Higher scores on this subscale indicate elevated stress levels.
Depression | Week 2
  The DASS also contains a depression subscale that enables us to assess depressive symptoms. Participants will provide responses related to their mood and emotional well-being, allowing us to gauge the extent of their depressive symptomatology. Higher scores on this subscale indicate a greater level of depressive symptoms.
Insomnia | Week 2
  The ISI consists of seven items that assess the severity of sleep-onset and sleep-maintenance difficulties, satisfaction with current sleep patterns, interference with daily functioning, noticeability of impairments attributed to sleep problems, and the level of distress caused by the sleep difficulties. Higher scores indicates greater insomnia severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Tecnocampus, Mataró, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No